CLINICAL TRIAL: NCT02965586
Title: Efficacy of Intrathecal Versus Intravenous Dexmedetomidine for Prevention of Post Spinal Anesthesia Shivering in Patients Undergoing TURP
Brief Title: Efficacy of Intrathecal Versus Intravenous Dexmedetomidine for Prevention of Post Spinal Anesthesia Shivering
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lecturer of anesthesia, ICU and pain managment, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 360
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Shivering
MeSH Terms: interventions — Injections, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- intravenous dexmedetomidine group (Active Comparator): intrathecal 2.5 ml of heavy bupivicaine 0.5% pulse 0.5 mg morphine and will receive intravenous dexmedetomidine infusion as prepared. Dexmedetomidine will be diluted to a volume of 50 ml (4 mg ml-1) and presented as coded syringes by an anesthesiologist. I.V. bolus of dexmedetomidine 1 ug kg-1 administered by a syringe pump over a 10-min period followed by an infusion of 0.4 ug kg-1h-1 dexmedetomidine during the surgery. Just after intrathecal injection, all drugs were infused intravenously. The infusions will be stopped at the end of surgery.
  Interventions: Drug: intrathecal
- intrathecal dexmedetomidine group (Active Comparator): intrathecal2.5 ml of heavy bupivicaine 0.5% pulse 0.5 mg morphine and dexmedetomidine (10µg) and will receive an equal volume of saline intravenously
  Interventions: Drug: intrathecal
- control group (Placebo Comparator): intrathecal 2.5 ml of heavy bupivicaine0.5% pulse 0.5 mg morphine and will receive an equal volume of saline intravenously
  Interventions: Drug: intrathecal

INTERVENTIONS:
Drug: intrathecal — intrathecal block will be performed in sitting position using 25 G spinal needle at either the L3-L4 or L4-L5 intervertebral spaces.

SUMMARY:
compare the efficacy of intrathecal versus intravenous dexmedetomidine in attenuation and prevention of shivering in TURP under spinal anesthesia in a randomized controlled trial.

DETAILED DESCRIPTION:
Shivering is a frequent complication following SA. It is distressing and unpleasant experience for patients. The incidence of shivering has been reported to be about 36-85% after SA. It is more common in TURP that may be due to absorption of large amount of irrigating fluid at room temperature. Shivering may occur as a response to hypothermia. However, it may also occur in normothermic patients. SA impairs the thermoregulation system by inhibiting tonic vasoconstriction below the level of anesthesia through sympathetic and somatic neural blockade. With internal redistribution of heat from the core to the peripheral compartment, the loss of thermoregulatory vasoconstriction results in increased heat loss from body surfaces in excess of metabolic heat production. Excessive shivering can result in an increased oxygen demand up to 400% of normal and induce metabolic derangements such as hypoxemia, lactic acidosis and hypercarbia. Therefore, shivering may cause problems in patients with low cardiac and pulmonary reserves.

Considering these undesirable consequences of shivering, measures to prevent in the postoperative period are important. Various drugs have been investigated for the prevention or treatment of postoperative shivering, including meperidine, ketamine, tramadol, doxapram and dexmedetomidine.

Dexmedetomidine is an α 2-agonist that decreases vasoconstriction and shivering thresholds and when administered with meperidine additively reduces the shivering threshold in healthy volunteers. Intraoperative dexmedetomidine reduces postanesthetic shivering as does meperidine after surgery.

One bolus dose of dexmedetomidine 1 μg/kg with or without continuous infusion was used in the previous antishivering studies. Dexmedetomidine also has sedative and analgesic effects in the postoperative period. Patients who received an intraoperative injection of dexmedetomidine were more sedated after surgery than those who received placebo. This can be a disadvantage particularly for patients undergoing outpatient surgery.

Addition of intrathecal dexmedetomidine to heavy bupivacaine 0.5% was more advantageous than fentanyl with special regard to its analgesic properties in diabetic surgical patients. Few studies have been done to evaluate the efficacy of intrathecal dexmedetomidine in attenuation and prevention of shivering in TURP.

We aimed to compare the efficacy of intrathecal versus intravenous dexmedetomidine in attenuation and prevention of shivering in TURP under spinal anesthesia in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo elective trans-urethral resection of the prostate(TURP) under spinal anesthesia.

Exclusion Criteria:

* Obese patients (BMI > 27)
* those with hypo- or hyperthyroidism,
* cardiopulmonary disease,
* psychological disorders,
* blood transfusion during surgery,
* Parkinsonians disease, and
* an initial body temperature above 38.0˚C or below 36.0 ˚C

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative shivering | 0, 10,20,30,40, 50,60 min
  Shivering will be assessed by Crossley and Mahajan scale where 0= No shivering, 1= Cyanosis and piloerection, 2 = Visible tremors only in one muscle group, 3 = Visible tremors in more than one muscle group, and 4 = intense shivering, tremors of the head, arm.

SECONDARY OUTCOMES:
sedation score | 0, 10,20, 30, 40, 50, 60 min
  a 5- point scale: 1 = fully awake and oriented, 2 = drowsy, 3 = eyes closed but open on command, 4 = eyes closed but open to mild physical stimulation, and 5 = eyes closed and unresponsive to mild physical stimulation
side effect | 0, 10,20, 30, 40, 50, 60 min
  hypotension, bradycardia, itching, nausea, vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Iorg0006563, Egypt

IPD SHARING:
Plan to Share IPD: No